CLINICAL TRIAL: NCT05923801
Title: Changing Tactics? Optimizing ECT in Difficult-to-treat Depression: A Randomized Trial Comparing Continuation of Right Unilateral ECT and Switching to Bitemporal ECT in Case of Early Non-response During an Acute Course of ECT for Difficult-to-treat Depression
Brief Title: Changing Tactics? Optimizing ECT in Difficult-to-treat Depression
Acronym: ChaT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Universiteit Antwerpen (Other); AZ Sint-Jan AV (Other); General Hospital Groeninge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S67329
Record Dates: First submitted 2023-06-01; First posted 2023-06-28 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Depression
Keywords: Electroconvulsive Therapy; Depression; Cognition
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Participants treated with ECT for depression, showing no 'response' (≥50 percent decrease in depressive symptom severity compared to baseline) after 4 treatment sessions will be randomized into 2 treatment groups: either continuation with RUL ECT or switch to BT ECT.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BT ECT (Active Comparator): Participants showing no response will be switched to BT ECT until remission is achieved.
  Interventions: Device: switch to BT electrode position
- RUL ECT (Active Comparator): Participants showing no response will continue with RUL ECT until remission is achieved.
  Interventions: Device: continue with RUL electrode position

INTERVENTIONS:
Device: switch to BT electrode position — use of different electrode positions of ECT device
  Arms: BT ECT
Device: continue with RUL electrode position — use of different electrode positions of ECT device
  Arms: RUL ECT

SUMMARY:
The goal of this randomized controlled trial is to address which treatment strategy (continue right unilateral (RUL) ECT or switch to bitemporal (BT) ECT speeds up recovery and has the least impact on memory function, in case of early non-response during an acute course of ECT for difficult-to-treat depression.

The main questions it aims to answer are:

* Assess the antidepressant efficacy and cognitive impact of the continuation of an ongoing treatment with RUL ECT compared to switching the treatment technique to BT ECT, in patients failing to show an early response to an acute course of ECT for major depression;
* Assess group and subject-specific trajectories of depressive symptom severity and neurocognitive performance during the acute ECT course and up to 3 months post-treatment.

Participants treated with ECT for depression, showing no 'response' (≥50 percent decrease in depressive symptom severity compared to baseline) after 4 treatment sessions, will be randomized to either switch to BT ECT or continue with RUL ECT. Mood and neurocognitive assessments will be performed at baseline, after 4 ECT sessions (before randomization), after 8 ECT sessions, at the end of the acute course and 3 month after the acute course.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
* Age 18 or older
* Diagnosis of major depressive disorder (DSM-5 296.21-30) or bipolar disorder, depressed (DSM-5 296.51-54; 296.84), confirmed by MINI (Mini International Neuropsychiatric Interview)

Exclusion Criteria:

* Contra-indication for general anesthesia
* Non-Dutch speaking
* Diagnosis of schizoaffective disorder or schizophrenia, confirmed by MINI
* Diagnosis of substance use disorder in the past six months, confirmed by MINI
* Diagnosis of neurocognitive disorder or intellectual disability alongside a MoCA score <23
* Previous ECT course in the past three months
* Participation in an interventional Trial with an investigational medicinal product or device
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change form baseline Depressive Symptom Severity | after 4 ECT sessions (2 weeks)
  mean scores on the Inventory of Depressive Symptomatology-Clinician Rated (IDS-CR)
Change form baseline Depressive Symptom Severity | after 8 ECT sessions (4 weeks)
  mean scores on the Inventory of Depressive Symptomatology-Clinician Rated (IDS-CR)
Depressive Symptom Severity | at the end of acute ECT course (up to 7 weeks)
  mean scores on the Inventory of Depressive Symptomatology-Clinician Rated (IDS-CR)
Depressive Symptom Severity | 3 months post-acute course
  mean scores on the Inventory of Depressive Symptomatology-Clinician Rated (IDS-CR)
Autobiographical Memory | after 4 ECT sessions (2 weeks)
  Mean scores on the Colombia University Autobiographical Memory Interview Short Form (CU-AMI-SF)
Autobiographical Memory | after 8 ECT sessions (4 weeks)
  Mean scores on the Colombia University Autobiographical Memory Interview Short Form (CU-AMI-SF)
Autobiographical Memory | at the end of acute ECT course (up to 7 weeks)
  Mean scores on the Colombia University Autobiographical Memory Interview Short Form (CU-AMI-SF)
Autobiographical Memory | 3 months post-acute course
  Mean scores on the Colombia University Autobiographical Memory Interview Short Form (CU-AMI-SF)

SECONDARY OUTCOMES:
Response/remission status | at the end of acute ECT course (up to 7 weeks)
  number of participants with an 50 percent decrease in IDS-score/ IDS-score < 12
number of ECT treatments needed to achieve response/remission | at the end of acute ECT course (up to 7 weeks)
Neurocognitive performance (RAVLT) | after 4 ECT sessions (2 weeks), after 8 ECT sessions (4 weeks), at the end of acute ECT course (up to 7 weeks), 3 months post-acute course
  mean scores on RAVLT (Rey Auditory Verbal Learning Test)
Neurocognitive performance (MoCA) | after 4 ECT sessions (2 weeks), after 8 ECT sessions (4 weeks), at the end of acute ECT course (up to 7 weeks), 3 months post-acute course
  mean scores on MoCA (Montreal Cognitive Assessment)
Neurocognitive performance (COWAT) | after 4 ECT sessions (2 weeks), after 8 ECT sessions (4 weeks), at the end of acute ECT course (up to 7 weeks), 3 months post-acute course
  mean scores on COWAT (Controlled Oral Word Association Test)
Neurocognitive performance (WMS-R) | after 4 ECT sessions (2 weeks), after 8 ECT sessions (4 weeks), at the end of acute ECT course (up to 7 weeks), 3 months post-acute course
  mean scores on WMS-R (Wechsler Memory Scale) (Cijferreeksen)

OTHER OUTCOMES:
Clinical characteristics (CORE) | after 4 ECT sessions (2 weeks), after 8 ECT sessions (4 weeks), at the end of acute ECT course (up to 7 weeks), 3 months post-acute course
  mean scores on CORE
Clinical characteristics (PDAS) | after 4 ECT sessions (2 weeks), after 8 ECT sessions (4 weeks), at the end of acute ECT course (up to 7 weeks), 3 months post-acute course
  mean scores on PDAS

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Sienaert, MD, PhD, Principal Investigator — UPC KU Leuven
Locations (1):
- UPC Kortenberg, Kortenberg, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Details on methodology are noted in the protocol. Questionnaires will be used as stated in their manuals. Data of assessments (informed consent, answers to questionnaires,...) are documented on paper and entered in a data platform (Redcap). When access is provided, or data is exported (using a certain standard format such as .xls or .cvs) it can be reused by other researchers. All data is provided with a clear nomenclature, referring to the scores of standardized questionnaires,cognitive assessment tools, ECT parameters,...
  Further, published articles by the involved researchers will contain all details necessary to reveal context of data collection, collection methodology, analytical and procedural information, etc.
  The pseudonymized data can be made available upon request, after permission is granted by the principal investigator and the head researchers.

REFERENCES:
- [Background] Kolshus E, Jelovac A, McLoughlin DM. Bitemporal v. high-dose right unilateral electroconvulsive therapy for depression: a systematic review and meta-analysis of randomized controlled trials. Psychol Med. 2017 Feb;47(3):518-530. doi: 10.1017/S0033291716002737. Epub 2016 Oct 26. PMID 27780482
- [Background] Semkovska M, Landau S, Dunne R, Kolshus E, Kavanagh A, Jelovac A, Noone M, Carton M, Lambe S, McHugh C, McLoughlin DM. Bitemporal Versus High-Dose Unilateral Twice-Weekly Electroconvulsive Therapy for Depression (EFFECT-Dep): A Pragmatic, Randomized, Non-Inferiority Trial. Am J Psychiatry. 2016 Apr 1;173(4):408-17. doi: 10.1176/appi.ajp.2015.15030372. Epub 2016 Feb 19. PMID 26892939
- [Background] Kellner CH, Knapp R, Husain MM, Rasmussen K, Sampson S, Cullum M, McClintock SM, Tobias KG, Martino C, Mueller M, Bailine SH, Fink M, Petrides G. Bifrontal, bitemporal and right unilateral electrode placement in ECT: randomised trial. Br J Psychiatry. 2010 Mar;196(3):226-34. doi: 10.1192/bjp.bp.109.066183. PMID 20194546
- [Background] Sackeim HA, Prudic J, Devanand DP, Nobler MS, Haskett RF, Mulsant BH, Rosenquist PB, McCall WV. The benefits and costs of changing treatment technique in electroconvulsive therapy due to insufficient improvement of a major depressive episode. Brain Stimul. 2020 Sep-Oct;13(5):1284-1295. doi: 10.1016/j.brs.2020.06.016. Epub 2020 Jun 22. PMID 32585354
- [Background] Lapidus KA, Kellner CH. When to switch from unilateral to bilateral electroconvulsive therapy. J ECT. 2011 Sep;27(3):244-6. doi: 10.1097/YCT.0b013e31820059e1. No abstract available. PMID 21681108
- [Background] Birkenhager TK, Roos J, Kamperman AM. Improvement after two sessions of electroconvulsive therapy predicts final remission in in-patients with major depression. Acta Psychiatr Scand. 2019 Sep;140(3):189-195. doi: 10.1111/acps.13054. Epub 2019 Jun 7. PMID 31104321
- [Background] Rush AJ, Gullion CM, Basco MR, Jarrett RB, Trivedi MH. The Inventory of Depressive Symptomatology (IDS): psychometric properties. Psychol Med. 1996 May;26(3):477-86. doi: 10.1017/s0033291700035558. PMID 8733206
- [Background] van Diermen L, van den Ameele S, Kamperman AM, Sabbe BCG, Vermeulen T, Schrijvers D, Birkenhager TK. Prediction of electroconvulsive therapy response and remission in major depression: meta-analysis. Br J Psychiatry. 2018 Feb;212(2):71-80. doi: 10.1192/bjp.2017.28. PMID 29436330
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Kirov G, Jauhar S, Sienaert P, Kellner CH, McLoughlin DM. Electroconvulsive therapy for depression: 80 years of progress. Br J Psychiatry. 2021 Nov;219(5):594-597. doi: 10.1192/bjp.2021.37. PMID 35048827
- [Background] Kellner CH, Obbels J, Sienaert P. When to consider electroconvulsive therapy (ECT). Acta Psychiatr Scand. 2020 Apr;141(4):304-315. doi: 10.1111/acps.13134. Epub 2019 Dec 23. PMID 31774547
- [Background] Kellner CH, Knapp RG, Petrides G, Rummans TA, Husain MM, Rasmussen K, Mueller M, Bernstein HJ, O'Connor K, Smith G, Biggs M, Bailine SH, Malur C, Yim E, McClintock S, Sampson S, Fink M. Continuation electroconvulsive therapy vs pharmacotherapy for relapse prevention in major depression: a multisite study from the Consortium for Research in Electroconvulsive Therapy (CORE). Arch Gen Psychiatry. 2006 Dec;63(12):1337-44. doi: 10.1001/archpsyc.63.12.1337. PMID 17146008
- [Background] Kellner CH, Husain MM, Knapp RG, McCall WV, Petrides G, Rudorfer MV, Young RC, Sampson S, McClintock SM, Mueller M, Prudic J, Greenberg RM, Weiner RD, Bailine SH, Rosenquist PB, Raza A, Kaliora S, Latoussakis V, Tobias KG, Briggs MC, Liebman LS, Geduldig ET, Teklehaimanot AA, Lisanby SH; CORE/PRIDE Work Group. Right Unilateral Ultrabrief Pulse ECT in Geriatric Depression: Phase 1 of the PRIDE Study. Am J Psychiatry. 2016 Nov 1;173(11):1101-1109. doi: 10.1176/appi.ajp.2016.15081101. Epub 2016 Jul 15. PMID 27418379
- [Background] Semkovska M, McLoughlin DM. Objective cognitive performance associated with electroconvulsive therapy for depression: a systematic review and meta-analysis. Biol Psychiatry. 2010 Sep 15;68(6):568-77. doi: 10.1016/j.biopsych.2010.06.009. Epub 2010 Jul 31. PMID 20673880
- [Background] Sackeim HA, Decina P, Kanzler M, Kerr B, Malitz S. Effects of electrode placement on the efficacy of titrated, low-dose ECT. Am J Psychiatry. 1987 Nov;144(11):1449-55. doi: 10.1176/ajp.144.11.1449. PMID 3314538
- [Background] Husain MM, Rush AJ, Fink M, Knapp R, Petrides G, Rummans T, Biggs MM, O'Connor K, Rasmussen K, Litle M, Zhao W, Bernstein HJ, Smith G, Mueller M, McClintock SM, Bailine SH, Kellner CH. Speed of response and remission in major depressive disorder with acute electroconvulsive therapy (ECT): a Consortium for Research in ECT (CORE) report. J Clin Psychiatry. 2004 Apr;65(4):485-91. doi: 10.4088/jcp.v65n0406. PMID 15119910
- [Background] Martinez-Amoros E, Goldberg X, Galvez V, de Arriba-Arnau A, Soria V, Menchon JM, Palao DJ, Urretavizcaya M, Cardoner N. Early improvement as a predictor of final remission in major depressive disorder: New insights in electroconvulsive therapy. J Affect Disord. 2018 Aug 1;235:169-175. doi: 10.1016/j.jad.2018.03.014. Epub 2018 Apr 6. PMID 29656263